CLINICAL TRIAL: NCT00454402
Title: Alfuzosin in Uretheric Stones
Brief Title: ALF-STONE: Alfuzosin in Uretheric Stones
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinued due to incomplete recruitment
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_9795; EudraCT # : 2005-005481-36
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alfuzosin

SUMMARY:
The aim of the study is to assess the effect of Alfuzosin compared with placebo, for 7 days, on the outcome of patients with uretheric stones submitted to Extracorporeal Shock Wave Lithotripsy (ESWL), namely in the percentage of patients without imagiologic evidence of any stone after 72h to 96 hours.

This study will also specifically focus on the evaluation of time of stone clearance and of pain reduction (Numeric Rating Scale).

ELIGIBILITY:
Inclusion criteria:

* Patients with imagiologic evidence of uretheric stones

Exclusion criteria:

* Women pregnant or breast feeding
* Patients with renal impairment (creatinine > 2mg/dl)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2006-08; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety: General clinical safety by collection of spontaneously reported adverse events | at each visit
Efficacy: Percentage of patients without imagiologic evidence of any stone | 72h to 96 hours after ESWL

SECONDARY OUTCOMES:
Percentage of patients without imagiologic evidence of any stone | 24 hours after ESWL
Percentage of patients with clinical evidence of stones clearance | 72h to 96 hours after ESWL
Time for stone clearance (clinical evaluation)
Numeric Rating Scale scores | at 24h, (48h, if applicable), 72-96h and 7 days
Need for rescue analgesic medication.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Santos, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Lisbon, Portugal